CLINICAL TRIAL: NCT03968510
Title: The Effect of Parathyroidectomy on Swallowing Related Quality of Life in Primary Hyperparathyroidism
Brief Title: Swalqol in Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Barış Sevinç, Assistant professor, Uşak University
Other Study IDs: pthswalqol
Record Dates: First submitted 2019-03-20; First posted 2019-05-30 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism | interventions — Parathyroidectomy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parathyroidectomy cases: patients who will be operated for primary hyperparathyroidism
  Interventions: Procedure: parathyroidectomy

INTERVENTIONS:
Procedure: parathyroidectomy — routine parathyroidectomy will be done for the treatment of adenoma

SUMMARY:
Swallow related quality of life before and after parathyroidectomy will be evaluated in patients with primary hyperparathyridism.

DETAILED DESCRIPTION:
Patients who will undergone parathyroidectomy for primary hyperparathyroidism will be included in the study. Swal-Qol and Sf-36 forms will be used for evaluation of quality of life before and 1 month after the surgery. The change in the quality of life and swallowing related quality of life will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* no diagnosis of Alzheimers disease
* must be able to swallow tablets Planned operation for primary hyperparathyroidism

Exclusion Criteria:

* secondary or tertiary hyperparathyroidism
* insulin dependent diabetes
* thyroid disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with primary hyperparathyroidism
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | 6 months
  Quality of life will be evaluated using short form 36

CONTACTS AND LOCATIONS:
Overall Officials: Barış Sevinç, Principal Investigator — Uşak University
Locations (1):
- Uşak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided